CLINICAL TRIAL: NCT01026012
Title: Maximal Bruce Protocol With the Use of Regadenoson For Myocardial Perfusion Stress Testing
Acronym: Rega Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Scott Jerome, Assistant Professor of Medicine, Director of Ambulatory Outreach Cardiology, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00040189
Record Dates: First submitted 2009-11-30; First posted 2009-12-04 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Function
Keywords: Regadenoson; 85% predicted heart rate; Myocardial perfusion stress testing
MeSH Terms: interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined Protocol (Experimental): patient with submaximal symptom limited maximal exercise testing will also be administered regadenoson pharmacological stress test.
  Interventions: Drug: regadenoson

INTERVENTIONS:
Drug: regadenoson — Regadenoson dose of 400 mcg will be infused over 10-20 seconds followed by a saline flush.

SUMMARY:
It is been known for at least 20 years that the hemodynamic data, the amount of exercise performed as well as symptoms on the treadmill, has significant value to the perfusion stress testing. When a pharmacologic stress test is performed (and adenosine stress test over 4-6 minutes), this hemodynamic data is lost. Because of this loss of valuable data, it is felt that there is also a loss of significant prognostic data as well. With the advent and FDA release of Regadenoson in a rapid injection form (over 10 seconds), it is thought that the combination of both exercise stress testing and pharmacologic testing in subjects that do not achieve 85% in a maximal predicted heart rate may be a viable stress testing option.

The purpose of this study is to look at using the drug, regadenoson, with exercise stress testing; and the side effect symptoms that may be experienced by individual subjects using this combination.

DETAILED DESCRIPTION:
A nuclear stress test has been recommended for a patient by their doctor. This test helps to detect significant blockages in the artery to the heart. The test involves the patient walking on a treadmill until their heart rate reaches 85% of their age-determined maximal predicted heart rate. If the patient needs to stop walking for any reason (tiredness, chest pain, shortness of breath or dizziness) prior to reaching the 85% of their maximal heart rate, then the test becomes inaccurate and blockages can be missed. Nonetheless, the information that we gain from the patient walking remains valuable.

If the subject does not reach 85%, the usual procedure is to re-do the test where the subject would not walk on the treadmill, but would be injected with a pharmacologic agent (drug) which dilates their blood vessels. This would allow us to obtain an accurate picture about any blockages in the blood vessels. By doing the "drug" test alone, we lose the important information gained by the treadmill test.

In the present study the subject will be asked to walk on the treadmill and near the end of the walk, if they do not reach 85%, then the "drug" will be given to the patient. Regadenoson is FDA approved for drug stress testing. Regadenoson (versus one of the other pharmacological agents) will be given at a dose of 400 mcg, will be infused over 10 - 20 seconds followed by standard flushing solution, and then the infusion of a radiotracer (the FDA approved method of administration) will be given for nuclear imaging. The entire intravenous procedure takes 30 seconds. The subject will then undergo 5 minutes of standard observation/monitoring post infusion administration. Standard nuclear stress imaging will then follow. By doing this, we will obtain all the important information from the exercise portion of this test and maintain the accuracy to detect blockages. By doing the study in this manner, we will be able to save the subject time and obtain more information about the heart than either test individually.

ELIGIBILITY:
Inclusion Criteria:

1. Referred for clinically indicated exercise stress Myocardial Perfusion Imaging (MPI) study, Provide written informed consent
2. Provide written informed consent

Exclusion Criteria:

1. Acute myocardial infarction or unstable angina within three months 2 Any condition judged by the investigator likely to pose a safety risk to the patient 3 Participation in another investigational drug study within one month, Or participation in any previous rate adenosine trial 4 Females who are breast-feeding or pregnant 5 Dipyridamole use within 48 hours 6 Consumption of methyl xanthine's, coffee theophylline, caffeinated soft drinks chocolate within 24 hours of the stress test 7 Has received a heart transplant 8 Has a recent history (less than 30 days) of uncontrolled ventricular arrythmia 9 Active respiratory wheezing, angina, ventricular dysrhythmia, low blood pressure or EKG changes 10 Patients that do not have a functioning artificial pacemaker and have either: 1) second or third degree atrialventicular block 2) sinus node dysfunction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Jerome, D.O., Principal Investigator — University of Maryland
Locations (1):
- University of MD Cardiology Physicians, Westminster, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period January 2010 to October 2010 occurred in outpatient office.
Groups:
- Combined Stress Group: Subjects had a sub-maximal symptom limited stress test (<85% MPHR)then immediately followed by pharmological stress test with the infusion of regadenoson 400mcg infused over 10-20 seconds.
Period: Overall Study
Arm/Group | Combined Stress Group
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Combined Stress Group: patient's were monitor for approximately 30 minutes following regadenoson infusion
Arm/Group | Combined Stress Group
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Side Effects, Including Dyspnea, Headache, Dizziness, Chest Pain, Nausea, Abdominal Discomfort, Dysgeusia, Flushing, and Symptomatic Hypotension and Others.
Description: Side effect will be monitored/reported by subject during stress test and 30 mins in recovery.( 1-2 hours total: for the during the subject was in the office for the test)
Time Frame: During and 30 minutes after stress test
Population: Subjects whom completed the combined stress test, including imaging
Measure: Number; unit: participants
Groups:
- Combined Stress Group: Side effect will be monitored/reported by subject during stress test and 30 mins in recovery.
Arm/Group | Combined Stress Group
Number analyzed (Participants) | 40
participants | 27

ADVERSE EVENTS:
Groups:
- Safety: patient's were monitor for approximately 30 minutes following regadenoson infusion
Arm/Group | Safety
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No